CLINICAL TRIAL: NCT06045065
Title: Establishment of Pre-clinical Stem Line and Tumoroid Models of Brain Tumors
Brief Title: Preclinical Brain Tumor Models
Acronym: HITCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM20_0037 - HITCH
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Brain Metastases; Diffuse Gliomas
Keywords: Brain metastases; Glioma; Glioblastoma; Preclinical models; Tumoroids; Cell lines
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fresh tumor sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with primitive tumor: Patient samples will be collected during routine care neurosurgical resection.
  Interventions: Other: Fresh tumor sampling
- patients with brain metastasis: Patient samples will be collected during routine care neurosurgical resection.
  Interventions: Other: Fresh tumor sampling

INTERVENTIONS:
Other: Fresh tumor sampling — Patient samples will be collected during neurosurgical resection. .

SUMMARY:
Background: Primary or secondary brain tumors (metastases) remain associated with a very poor prognosis linked to significant therapeutic resistance. Thus, glioblastoma, which is the most common and aggressive primary brain tumor in adults, is associated with inevitable relapses within 7 to 10 months and median survival of approximately 12 to 14 months. At the same time, brain metastases are increasingly increasing following better systemic control of other metastatic sites and improvement in detection methods. However, they remain resistant to the latest therapeutic innovations such as immunotherapies or targeted therapies.

In this context, innovative strategies are necessary to identify new therapeutic targets and implement new treatments to overcome resistance phenomena in the clinic.

Objective: Our goal will be to generate tumoroids and stem-like cell lines (PDX) from patient tumor samples.

Methods: We will establish tumor tumoroids and stem cell lines from patient samples. These preclinical models will allow us to test a large number of drugs, quickly and efficiently thanks to models as close as possible to patient tumors and limiting the use of animal models (3R).

Overall, this project should enable major advances in the treatment of glioblastoma and brain metastases and enable the rapid testing of new molecules in clinical trials thanks to the homology of our models with our patients' diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Brain tumor neuro-imaging
* Eligible for neurosurgery

Exclusion Criteria:

* unresectable tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with primitive tumor or with brain metastasis
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Tumoroid and stem cell line generation | 4 weeks after generation
  The generation of tumoroids and stem cell lines will be attested at 4 weeks after initiation of their culture.
  Tumoroids: generation of round and viable structures Stem cell lines: generation of neurospheres

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance publique hopitaux de marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No